CLINICAL TRIAL: NCT01310920
Title: The Role of Angiotensinogen Gene Polymorphism in the Pathogenesis of Non-familial Sick Sinus Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Jan-Yow Chen, China Medical University hospital
Other Study IDs: DMR99-IRB-316
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Sick Sinus Syndrome
MeSH Terms: conditions — Sick Sinus Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (2):
- sick sinus syndrome
  Interventions: Other: observation
- control

INTERVENTIONS:
Other: observation — genotyping
  Groups: sick sinus syndrome

SUMMARY:
Evidence has been documented for the close relationship between the arrhythmia pathogenesis and the gene expression in renin-angiotensin system. However, it remains unclear for involvement of RAS in the pathogenesis of non-familial sick sinus syndrome. The researchers thus investigated the possible relationship between non-familial sick sinus syndrome and the polymorphism and haplotype of the AGT promoter.

ELIGIBILITY:
Inclusion Criteria:

* sick sinus syndrome

Exclusion Criteria:

* 1.Severe systemic disease.
* 2.Acute coronary syndrome.
* 3.bradycardia with reversible cause.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The case group includes 200 patients and the control group includes 200 patients.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Yow Chen, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Dawan, Taiwan, Taiwan

REFERENCES:
- [Background] Mangrum JM, DiMarco JP. The evaluation and management of bradycardia. N Engl J Med. 2000 Mar 9;342(10):703-9. doi: 10.1056/NEJM200003093421006. No abstract available. PMID 10706901